CLINICAL TRIAL: NCT06640387
Title: CARE-ID: Dynamics of Respiratory Infections in Children and Transmission in Households and Schools
Status: Recruiting | Type: Observational
Sponsor: The Hospital for Sick Children (Other)
Responsible Party: Principal Investigator, Michelle Science, Staff Physician, The Hospital for Sick Children
Other Study IDs: 1000081729
Record Dates: First submitted 2024-10-10; First posted 2024-10-15 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: SARS CoV 2 Infection; RSV Infection; Influenza; Mycoplasma Pneumoniae; Bordetella Pertussis, Whooping Cough
MeSH Terms: conditions — COVID-19; Respiratory Syncytial Virus Infections; Influenza, Human; Whooping Cough

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Respiratory samples (e.g. saliva, nasal, nasopharyngeal specimens) for future respiratory infection testing (no human genetic testing)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Daily Influenza, RSV or SARS-CoV-2 PCR testing for 14 days — Each participant will undergo daily PCR testing for Influenza, RSV or SARS-CoV-2 to assess viral dynamics

SUMMARY:
Viral respiratory tract infections are very common in children. They contribute to missed time in school, work disruption for caregivers and can also cause severe illness requiring hospitalization and rarely death. In the 2022-2023, influenza, RSV and SARS-CoV-2 viruses infected a large number of children which strained the pediatric healthcare system in many jurisdictions. Unfortunately, there continues to be limited data on duration of infectiousness and transmission risk of these viruses to inform public health decisions during times when there is significant circulation of these viruses.

ELIGIBILITY:
Inclusion Criteria:

Viral dynamics (primary outcome):

* The child must be less than 18 years of age
* Have a positive PCR sample for influenza, RSV or SARS-CoV-2,
* Have any one of the symptoms listed to meet testing eligibility: fever, cough, shortness of breath, decreased or loss of taste or smell, muscle aches/joint pains (unusual, long lasting, not related to injury), extreme tiredness (unusual fatigue not otherwise explained), sore throat, runny or stuffy/congested nose, headache (new, unusual, long-lasting), nausea/vomiting and/or diarrhea, and
* Be within 5 days of symptom onset

Household testing inclusion criteria (secondary outcome):

-Any individual in the same household (i.e. household contacts, defined as residing at the same address) as the individual testing positive by PCR for influenza, RSV, SARS-CoV-2, mycoplasma pneumoniae, or bordetella pertussis

Classroom testing inclusion criteria (secondary outcome):

-Any individual in the same classroom (i.e. classroom contacts) as the individual testing positive by PCR for influenza, RSV, SARS-CoV-2, mycoplasma pneumoniae, or bordetella pertussis (i.e. case identified through the THS program)

Exclusion Criteria:

Viral dynamics (primary outcome):

-Participants will be ineligible if they are more than 5 days from symptom onset

Min Age: 1 Day | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Individuals with acute symptomatic influenza, RSV, SARS-CoV-2, mycoplasma pneumoniae, or bordetella pertussis infection identified through hospital testing (inpatient, outpatient, staff household members) or the school-based take-home saliva testing program.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2024-10-10 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
To describe the viral dynamics of influenza, RSV and SARS-CoV-2 over time among children <18 years of age. | 14 days
  The correlation between symptom onset and symptom resolution and viral load for each virus will be described.

SECONDARY OUTCOMES:
To assess the impact of various host factors on viral dynamics | 14 days
  The correlation between host factors and viral dynamics will be explored.
To assess the frequency of influenza, RSV, SARS-CoV-2, mycoplasma pneumoniae and bordetella pertussis transmission in households. | Within 14 days of case identification
  The number of household contacts that are tested and test positive for the same respiratory virus (influenza, RSV, SARS-CoV-2, mycoplasma pneumoniae, bordetella pertussis) will be described.
To examine the risk factors for influenza, RSV, SARS-CoV-2, mycoplasma pneumoniae and bordetella pertussis transmission in households | Within 14 days of case identification
  The correlation between household characteristics and transmission of each of the viruses will be explored.
To assess the frequency of influenza, RSV, SARS-CoV-2, mycoplasma pneumoniae and bordetella pertussis transmission in classrooms. | Within 14 days of case identification
  The number of classmates in the classroom that are tested and test positive for the same respiratory virus (influenza, RSV, SARS-CoV-2, mycoplasma pneumoniae, bordetella pertussis) will be described.
To examine the risk factors for influenza, RSV, SARS-CoV-2, mycoplasma pneumoniae and bordetella pertussis transmission in classrooms | Within 14 days of case identification
  The correlation between classroom characteristics and transmission of each virus in classrooms will be explored.

CONTACTS AND LOCATIONS:
Overall Officials: Michelle Science, Principal Investigator — The Hospital for Sick Children (SickKids)
Locations (1):
- The Hospital for Sick Children (SickKids), Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
Data elements will be made available by request with appropriate documentation and approvals.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data will be made available once the study is complete and published.
Access Criteria: upon request with appropriate approvals